CLINICAL TRIAL: NCT02961140
Title: The Effects of Different Anesthetic Managements on Inflammation, Oxidative Injuries, and Major Organ Complications: a Prospective Investigations on Esophageal Reconstruction and Intraoperative Shock
Brief Title: Different Anesthetic Managements of Esophageal Resection and Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201512052RINB
Record Dates: First submitted 2016-11-06; First posted 2016-11-10 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Anesthesia; Esophagus Cancer; Postoperative Complications
Keywords: Outcome
MeSH Terms: conditions — Esophageal Neoplasms; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardiac Output Maximization (Experimental): maximize stroke volume, and maintain cardiac index and stroke volume variation during the whole operation
  Interventions: Other: Cardiac Output Maximization
- Cardiac Output Normalization (Active Comparator): keep cardiac index (CI) ≥ 2.2, and maintain CI and stroke volume variation during the whole operation
  Interventions: Other: Cardiac Output Normalization

INTERVENTIONS:
Other: Cardiac Output Maximization — According to Frank-Starling law, the investigator will administer Voluven 6% 250 mL every 5 minute until stroke volume maximized (stabilized for 20 minutes), and maintain cardiac index and stroke volume variation during the whole operation.
  Arms: Cardiac Output Maximization
Other: Cardiac Output Normalization — The investigator will administer intravenous fluids to keep cardiac index (CI) ≥ 2.2, and maintain CI and stroke volume variation during the whole operation.
  Arms: Cardiac Output Normalization

SUMMARY:
Anesthetic management and fluid therapy is crucial in esophageal resection and reconstruction, which is associated with high incidence of postoperative morbidity and mortality. This study aims to investigate the effect of goal directed fluid management on the postoperative outcome of esophageal resection and reconstruction.

DETAILED DESCRIPTION:
Anesthetic management and fluid therapy is crucial in esophageal resection and reconstruction, which is associated with high incidence of postoperative morbidity and mortality. Excessive fluid administration may result in pulmonary complication, while extremely hypovolemia may lead to shock, circulatory dysfunction, and renal damage. Little is known about fluid status will have impact on anastomotic leakage. Goal-directed fluid therapy has shown to benefit perioperative outcome in major abdominal surgery. This study aims to investigate the effect of goal directed fluid management on the postoperative outcome of esophageal resection and reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as esophageal cancer
* Scheduled for minimally invasive esophageal resection and reconstruction

Exclusion Criteria:

* End-stage organ dysfunction, including heart failure, hepatic failure, renal failure
* Arrhythmia
* Pregnancy

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative complication | 1 month
  Perioperative mortality, anastomotic leakage, pneumonia, respiratory failure, renal dysfunction, and surgical site infection

SECONDARY OUTCOMES:
Intraoperative hemodynamic stability | 1 day
  Incidence of intraoperative shock, use of vasopressor or inotropic agents
Length of stay | 1 month
  Intensive care unit length of stay and hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Ya-jung Cheng, M.D., Ph.D, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No